CLINICAL TRIAL: NCT01746147
Title: Assessment of Body, Liver and Labile Plasma Iron and Their Association With Outcome and Immunological Recovery in MDS or AML Patients Undergoing Allogeneic Stem Cell Transplantation - ALLIVE (ALLogeneic Iron inVEstigators) Observational Trial
Brief Title: Assessment of Body, Liver and Labile Plasma Iron and Their Association With Outcome and Immunological Recovery in Myelodysplastic Syndrome (MDS) or Acute Myeloid Leukemia (AML) Patients Undergoing Allogeneic Stem Cell Transplantation - ALLIVE (ALLogeneic Iron inVEstigators) Observational Trial
Acronym: ALLIVE
Status: Completed | Type: Observational
Sponsor: GWT-TUD GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: ALLIVE-2012
Record Dates: First submitted 2012-12-05; First posted 2012-12-10 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: MDS and AML Prior to Allogeneic SCT
Keywords: MDS; AML; allogeneic SCT
MeSH Terms: interventions — Pharmaceutical Preparations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with MDS and AML prior to allogeneic SCT
  Interventions: Other: No intervention and study treatment

INTERVENTIONS:
Other: No intervention and study treatment

SUMMARY:
The ALLIVE (ALLogeneic Iron inVEstigators) trial aims at quantifying the extent and dynamic change of LPI occurrence during conditioning and at identifying LPI-predictive peri-transplant parameters. Further points of interest are the improvement of systemic iron overload (SIO) diagnostics and the correlation of different SIO parameters with outcome after transplantation. The results of this trial will help to design prospective interventional studies addressing therapeutic options in patients at risk for SIO-associated toxicity during allogeneic stem-cell transplantation (allo-SCT).

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years at the time of signing the informed consent form
* Signed informed consent
* Diagnosis of AML or MDS according to WHO classification
* Planned allogeneic stem cell transplantation after reduced intensity or myeloablative conditioning from related or unrelated donors
* At risk for iron toxicity as defined by ferritin >500 ng/ml and/or history of more than 10 RBC transfusions prior to allo-SCT

Exclusion Criteria:

* Claustrophobia or other mental disorders making MRI imaging unbearable for the patient
* Cardiac pacemakers, metal implants splinters or other contraindications for MRI
* More than 1 Human leukocyte antigen (HLA) allele or antigen mismatch between donor and recipient
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Patients with a history of chronic drug abuse or another illness which does not allow the patient to assess the nature and/or possible consequences of the study
* Patients who are not likely to follow the trial protocol (lack of willingness to cooperate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women with AML or MDS according to WHO classification.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2012-12; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Description of dynamic changes of LPI prior, during and after conditioning for allo-SCT using standard descriptive parameters (Mean or Median and appropriate confidence intervals) | one year

SECONDARY OUTCOMES:
• Correlation coefficient of Liver iron concentration (LIC) and duration of detectable LPI during and after conditioning | one year
• Area under the Receiver-Operator-Characteristic (ROC) as well as sensitivity and specificity of specific thresholds of serum ferritin and transfusion history for prediction of LIC | one year
• Association of serum ferritin and LIC with hematopoietic cell transplantation comorbidity index (HCT-CI) | one year
• Time course of LPI, enhanced labile plasma iron (eLPI), directly chelatable iron (DCI) and hepcidin during allo-SCT | one year
• Association of detectable LPI or eLPI during conditioning and occurrence of elevated liver enzymes during in hospital treatment course for allo-SCT | one year
• Cumulative incidence of graft versus host disease (aGvHD) grade 2-4 with respect to serum ferritin >1000 µg/l, transfusion burden >20 units of Red blood cells (RBC), LIC >125 µmol/g, peak value and duration of detectable labile plasma iron above median | one year
• Cumulative incidence of day 100 non-relapse mortality (NRM) with respect to serum ferritin >1000 µg/l, transfusion burden >20 units of RBC, LIC >125 µmol/g and peak value and duration of detectable labile plasma iron above median | one year
• Cumulative incidence of infections with respect to serum ferritin >1000 µg/l, transfusion burden >20 parasitized red blood cell (PRBC), LIC >125 µmol/g and peak value and duration of detectable labile plasma iron above median | one year
• Median change of serum ferritin and LIC 100 days and 1 year after allo-SCT | one year
• Association between immune profile and iron parameters (serum ferritin >1000 µg/l, transfusion burden >20 units RBC, LIC >90 µmol/g and peak value and duration of detectable labile plasma iron above median | one year

CONTACTS AND LOCATIONS:
Overall Officials: Martin Wemke, MD, Principal Investigator — on behalf of GWT
Locations (5):
- Germany (5):
  - III. Medizinischen Klinik Hämatologie und Internistische Onkologie Universitätsmedizin Mannheim, Mannheim, Baden-Wurttemberg
  - III. Medizinischen Klinik des Klinikums rechts der Isar, München, Bavaria
  - Universitätsklinikum MKII, Hämatologie/Onkologie, Universitäres Zentrum für Tumorerkrankungen, Frankfurt am Main, Hesse
  - Medizinische Klinik und Poliklinik III Abteilung für Hämatologie und Onkologie Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Carl Gustav Carus der TU Dresden Medizinische Klinik und Poliklinik I, Dresden, Saxony

REFERENCES:
- [Derived] Wermke M, Eckoldt J, Gotze KS, Klein SA, Bug G, de Wreede LC, Kramer M, Stolzel F, von Bonin M, Schetelig J, Laniado M, Plodeck V, Hofmann WK, Ehninger G, Bornhauser M, Wolf D, Theurl I, Platzbecker U. Enhanced labile plasma iron and outcome in acute myeloid leukaemia and myelodysplastic syndrome after allogeneic haemopoietic cell transplantation (ALLIVE): a prospective, multicentre, observational trial. Lancet Haematol. 2018 May;5(5):e201-e210. doi: 10.1016/S2352-3026(18)30036-X. Epub 2018 Apr 5. PMID 29628397